CLINICAL TRIAL: NCT05940116
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-20117 in Participants With Advanced Solid Tumors
Brief Title: A Phase I Clinical Study of HS-20117 in Participants With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20117-101
Record Dates: First submitted 2023-06-26; First posted 2023-07-11 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Non-Small Cell Lung Cancer; Solid Tumor
Keywords: Non-Small Cell Lung Cancer; Solid Tumor; HS-20117; Epidermal Growth Factor Receptor; c-Mesenchymal-Epithelial Transition; Bispecific Antibody; EGFR exon 20 insertion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-20117 (Experimental): Participants will receive IV infusion of HS-20117 once during cycle 1 and once every 2 weeks during subsequent cycles (The duration of each treatment cycle is 28 days)
  Interventions: Drug: HS-20117

INTERVENTIONS:
Drug: HS-20117 — Phase Ia: patients will receive HS-20117 starting at 400 mg, and subsequent cohorts will test escalating doses, if tolerated, until a maximum tolerated dose (MTD) or maximum applicable dose (MAD) is defined.
  Phase Ib: patients will receive HS-20117 at MED or MAD
  Other Names: PM1080

SUMMARY:
HS-20117 is a fully-human EGFR-MET immunoglobulin G1(IgG1)-like bispecific antibody. The purpose of study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of HS-20117 as a monotherapy for participants with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase I clinical study of HS-20117 to evaluate the safety, tolerability, PK, immunogenicity and efficacy in participants with advanced solid tumors. The study consists of phase Ia (dose escalation) and phase Ib (dose expansion). The dose-escalation study will be performed to evaluate the safety, tolerability, PK profile, immunogenicity, and efficacy of HS-20117 in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) mutations. The subsequent dose-expansion study will be performed to evaluate the efficacy of HS-20117 in participants with locally advanced or metastatic NSCLC who have progressed after prior platinum-based chemotherapy or are intolerant to platinum-based chemotherapy with EGFR exon 20 insertion mutations, and to explore the efficacy of HS-20117 in participants with other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 - 75 years (inclusive).
2. For the phase Ia study: Participants with locally advanced or metastatic NSCLC (stage IIIB/IIIC/IV) with EGFR-activating mutations who have progressed after or are intolerant to or not available to standard of care (SoC).
3. For the phase Ib study:

   Cohort A: Participants with locally advanced or metastatic NSCLC (stage IIIB/IIIC/IV) with EGFR exon 20ins mutations who have progressed after prior platinum-based chemotherapy or are intolerant to platinum-based chemotherapy.

   Cohort B: Participants with other advanced solid tumors who have progressed after prior SoC or are intolerant to SoC.
4. Agree to provide fresh or archival tumor tissue.
5. At least one target lesion per the RECIST v1.1.
6. ECOG performance status of 0-1.
7. Minimum life expectancy > 12 weeks.
8. Males or Females should be using adequate contraceptive measures throughout the study.
9. Females must not be pregnant at screening or have evidence of non-childbearing potential.
10. Have signed Informed Consent Form.

Exclusion Criteria:

1. Received or are receiving the following treatments:

   1. For the phase Ib study Cohort A: Previous or current treatment with EGFR exon 20ins targeted therapy.
   2. Traditional Chinese medicine indicated for tumors within 2 weeks prior to the first dose of HS-20117.
   3. Cytotoxic chemotherapies, investigational drugs or other systematic anti-tumor therapies within 3 weeks prior to the first dose of HS-20117.
   4. Antibodies within 4 weeks prior to the first dose of HS-20117.
   5. Local radiotherapy within 2 weeks prior to the first dose of HS-20117, more than 30% of bone marrow irradiation or large-area radiotherapy within 4 weeks before the first dose of HS-20117.
   6. Presence of pleural effusion/ascites requiring clinical intervention; presence of pericardial effusion.
   7. Major surgery within 4 weeks prior to the first dose of HS-20117.
2. Presence of Grade ≥ 2 toxicities due to prior anti-tumor therapy.
3. History of other primary malignancies.
4. Untreated, or active central nervous system metastases.
5. Inadequate bone marrow reserve or organ functions.
6. Severe, uncontrolled or active cardiovascular disorders.
7. Severe or uncontrolled systemic diseases.
8. Severe bleeding symptoms or bleeding tendencies within 1 month prior to the first dose of HS-20117.
9. Severe arteriovenous thrombosis occurred within 3 months prior to the first dose of HS-20117
10. Serious infection within 4 weeks prior to the first dose of HS-20117.
11. Active infectious diseases.
12. Interstitial lung disease (ILD).
13. Serious neurological or mental disorders.
14. History of hypersensitivity to any component of HS-20117 or similar drugs.
15. Participants with any condition that compromises the safety of the participant or interferes with the assessment of the study, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
[Phase 1a] Maximum tolerated dose (MTD) of HS-20117 | Cycle 1 (28 days)
  MTD is defined as the previous dose level at which 2 or more out of 2-6 subjects experienced a DLT.
[Phase 1a] Maximum applicable dose (MAD) of HS-20117 | Cycle 1 (28 days)
  MAD is defined as follows: a) based on PK data, it is anticipated that at this dose level, the dose-exposure plateau has been reached, b) based on existing safety data, it is judged that dose escalation following this dose level will have a large safety risk or subject intolerance, or c) based on the PK-PD model, it suggested that the optimal target concentration of safety and efficacy has been explored.
[Phase 1b] Efficacy of HS-20117: Objective response rate (ORR) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  ORR is defined as the percentage of participants with BOR of confirmed CR or confirmed PR per RECIST v1.1

SECONDARY OUTCOMES:
[phase 1a and 1b] Incidence and severity of treatment-emergent adverse events | From the date of first dose until 90 days after the final dose. A cycle is 28 days
  Adverse event (assessed according to NCI CTCAE v5.0) is defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
[phase 1a and 1b] PK parameters: Maximum serum concentration (Cmax) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days.
  The Cmax is the maximum observed serum concentration of HS-20117.
[phase 1a and 1b] PK parameters: Trough serum concentration (Ctrough) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days.
  Ctrough is the observed serum concentration immediately prior to the next administration.
[phase 1a and 1b] PK parameters: Time to reach maximum observed serum concentration (Tmax) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days
  The Tmax is defined as time to reach maximum observed serum concentration of HS-20117.
[phase 1a] PK parameters: Area under the curve from time Zero to end of dosing interval (AUCtau) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days.
  The AUCtau is defined as the area under the serum concentration-time curve during a dose interval time period (tau).
[phase 1a] PK parameters: Terminal elimination half-life (t1/2) of HS-20117 | From the date of first dose until 30 days after the final dose. A cycle is 28 days.
  The t1/2 is defined as the time it takes for the concentration levels to fall to 50% of their value.
[phase 1a] Efficacy of HS-20117: ORR | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years.
  ORR is defined as the percentage of participants with BOR of confirmed CR or confirmed PR per RECIST v1.1.
[phase 1a and 1b] Efficacy of HS-20117: disease control rate (DCR) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years.
  DCR is deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 6 weeks) per RECIST v1.1.
[phase 1a and 1b] Efficacy of HS-20117: duration of response (DoR) | From the date of CR, PR until the date of disease progression or death, approximately 2 years.
  DoR only applies to participants whose best overall response is CR or PR based on assessment per RECIST v1.1. The start date is the date of first documented response of CR or PR (i.e. the start date of observed response, not the date when response was confirmed), and the end date is defined as the date of the first documented progression or death due to underlying disease.
[phase 1a and 1b] Efficacy of HS-20117: progression free survival (PFS) | From the date of randomization or first dose (if randomization is not needed) until the date of disease progression or death, approximately 2 years.
  PFS is defined as the time from the date of randomization or first dose (if randomization is not needed) to the date of the first documented progression or death due to any cause. PFS will be assessed per RECIST v1.1.
[phase 1b] Efficacy of HS-20117: overall survival (OS) | From the date of randomization or first dose (if randomization is not needed) until the documentation of death from any cause, approximately 4 years
  OS is defined as the time from the date of randomization or first dose (if randomization is not needed) to the date of death due to any cause. For each participant who is not known to have died as of the cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
[phase 1a and 1b] Immunogenicity of HS-20117 | Cycle 1 Day 1: predose through EOT or follow up period (90 days after the last dose).
  Immunogenicity will be measured by the number of participants that are ADA positive.

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China